CLINICAL TRIAL: NCT03150329
Title: A Phase 1 Study of Pembrolizumab Plus Vorinostat for Relapsed or Refractory Diffuse Large B-Cell Lymphoma, Follicular Lymphoma, and Hodgkin Lymphoma
Brief Title: Pembrolizumab and Vorinostat in Patients With Relapsed or Refractory DLBCL, FCL or HL.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17080; NCI-2017-00800 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17080 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Grade 3b Follicular Lymphoma; Recurrent B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between DLBCL and Classic HL; Recurrent Classic Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Refractory B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between DLBCL and Classic HL; Refractory Classic Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Refractory Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — pembrolizumab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vorinostat 100mg + Pembrolizumab 200mg (Experimental): Patients receive Vorinostat 100mg PO BID on days 1-5 and 8-12 and pembrolizumab 200mg IV over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Vorinostat
- Vorinostat 200mg + Pembrolizumab 200mg (Experimental): Patients receive Vorinostat 200mg PO BID on days 1-5 and 8-12 and pembrolizumab 200mg IV over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Vorinostat

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I trial studies the side effects and best dose of vorinostat when given together with pembrolizumab in treating patients with diffuse large B-cell lymphoma, follicular lymphoma, or Hodgkin lymphoma that has come back after a period of improvement or that does not respond to treatment. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer and may interfere with the ability of cancer cells to grow and spread. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving vorinostat and pembrolizumab together may work better than pembrolizumab alone in treating patients with diffuse large B-cell lymphoma, follicular lymphoma, or Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of vorinostat plus pembrolizumab therapy by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

II. To determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of vorinostat when given in combination with pembrolizumab.

SECONDARY OBJECTIVE:

I. To obtain preliminary estimates of the anti-tumor activity of pembrolizumab plus vorinostat therapy by assessing the overall response rate (ORR), complete response (CR) rate, duration of response (DOR), overall survival (OS) and progression-free survival (PFS).

EXPLORATORY OBJECTIVES:

I. Evaluate responses and disease progression according to the Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC).

II. Explore genomic biomarkers of response and resistance to pembrolizumab plus vorinostat therapy in patients with diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), or Hodgkin lymphoma (HL).

III. Explore immunologic biomarkers of response and resistance to pembrolizumab plus vorinostat therapy in patients with DLBCL, FL, or HL.

IV. Explore the value of circulating deoxyribonucleic acid (DNA) (ctDNA) as a biomarker of response to pembrolizumab plus vorinostat therapy.

OUTLINE: This is a dose-escalation study of vorinostat.

Patients receive vorinostat orally (PO) twice daily (BID) on days 1-5 and 8-12 and pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of follicular lymphoma, diffuse large B-cell lymphoma, or classical Hodgkin lymphoma according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution

  * FL: grade 1, 2, 3A, or 3B are eligible
  * DBLCL: transformed indolent lymphomas (TIL), primary mediastinal large B-cell lymphoma (PMBCL), and aggressive B-cell lymphoma unclassified (BCL-U) are eligible
  * HL: all classical HL subtypes are eligible except for nodular lymphocyte predominant Hodgkin lymphoma, which is excluded
* Patients with HL or DLBCL must refuse or not be candidates for curative autologous stem cell transplantation
* Have relapsed or refractory disease after at least 1 prior regimen, including:

  * Recurrence of disease after a documented complete response (CR)
  * Progression of disease after a partial response (PR) to the prior regimen
  * Partial response (PR), stable disease (SD) or progressive disease (PD) at the completion of the prior treatment regimen; if a patient has PR to prior regimen without PD, there must be biopsy-proven residual disease that is measurable
* Documented informed consent of the participant or legally authorized representative
* Have measurable disease by computed tomography (CT) or positron emission tomography (PET) scan, with one or more sites of disease >= 1.5 cm in longest dimension
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion prior to starting study therapy or from archival tissue of a biopsy that was performed after the most recent systemic therapy
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,000/mcL (within 14 days of treatment initiation)
* Platelets >= 75,000/mcL (within 14 days of treatment initiation)
* Hemoglobin >= 8 g/dL without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment (within 14 days of treatment initiation)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance (CrCl) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (within 14 days of treatment initiation)
* Serum total bilirubin =< 1.5 x ULN or =< 3 x ULN if patient has Gilberts disease OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 14 days of treatment initiation)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver involvement by lymphoma as the etiology of transaminase elevation (within 14 days of treatment initiation)
* Albumin >= 2.5 mg/dL (within 14 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 14 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 14 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication; Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy; Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has received a prior allogeneic hematopoietic stem cell transplant within the past 5 years, requires immunosuppression, or has evidence of active graft-versus-host-disease
* Has received prior autologous hematopoietic stem cell transplant within the last 60 days
* Has a known history of active TB (Bacillus tuberculosis)
* Severe hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 3 weeks earlier; if a patient has progressive or stable disease to prior regimen, rituximab is allowed up to 2 weeks prior to the initiation of study therapy
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study; Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has taken valproic acid, or another histone deacetylase inhibitor, within 2 weeks prior to study day 1
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement; subjects with prior CNS involvement by lymphoma must have remission of the CNS component of the lymphoma; these subjects must have a baseline magnetic resonance imaging (MRI) during screening without evidence of new or enlarging brain lesions and must not have any new or progressive neurologic symptoms
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; a history of hemolytic anemia associated with the lymphoma does not exclude a patient from the study
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a QT interval corrected for heart rate (QTc) > 470 ms using the Fridericia formula; if the screening electrocardiogram (ECG) has a QTc > 470ms, the mean QTc of 3 electrocardiograms (ECGs) can be utilized, but must be < 470 ms
* Is unable to swallow capsules, has a partial or small bowel obstruction, or has a gastrointestinal condition resulting in a malabsorptive syndrome (e.g. small bowel resection with malabsorption)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy; Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2026-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Godfrey J, Mei M, Chen L, Song JY, Bedell V, Budde E, Armenian S, Puverel S, Nikolaenko L, Chen R, Daniels S, Kennedy N, Peters L, Rosen ST, Forman SJ, Popplewell LL, Kwak LW, Herrera AF. Results from a phase I trial of pembrolizumab plus vorinostat in relapsed/refractory B-cell non-Hodgkin lymphoma. Haematologica. 2024 Feb 1;109(2):533-542. doi: 10.3324/haematol.2023.283002. PMID 37470137
- [Derived] Mei M, Chen L, Godfrey J, Song J, Egelston C, Puverel S, Budde LE, Armenian S, Nikolaenko L, Nwangwu M, Guo W, Gao L, Lee P, Chen R, Daniels S, Kennedy N, Peters L, Zain J, Rosen S, Forman S, Popplewell L, Kwak L, Herrera AF. Pembrolizumab plus vorinostat induces responses in patients with Hodgkin lymphoma refractory to prior PD-1 blockade. Blood. 2023 Oct 19;142(16):1359-1370. doi: 10.1182/blood.2023020485. PMID 37339586

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vorinostat 100mg + Pembrolizumab 200mg | Vorinostat 200mg + Pembrolizumab 200mg
Started | 6 | 46
Completed | 6 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat 100mg + Pembrolizumab 200mg | Vorinostat 200mg + Pembrolizumab 200mg | Total
Number analyzed (Participants) | 6 | 46 | 52
Age, Continuous [Median (Full Range); unit: years] | 53 [27 to 78] | 39 [18 to 79] | 40 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 16 | 17
  Male | 5 | 30 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 4 | 35 | 39
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 5 | 31 | 36
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 46 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade 3-5 Adverse Events
Description: Adverse events were assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From initial study treatment to 90 days post-last dose, up to 27 months.
Measure: Number; unit: participants
Arm/Group | Vorinostat 100mg + Pembrolizumab 200mg | Vorinostat 200mg + Pembrolizumab 200mg
Number analyzed (Participants) | 6 | 46
participants | 3 | 28

2. Primary Outcome: Maximum Tolerated Dose (MTD) on Vorinostat
Description: MTD is defined as the highest dose level at which < 33% of evaluable subjects experienced DLT, when at least 6 patients were treated at that dose level. The MTD was considered the recommended phase II dose (RP2D), however the principal investigator may ultimately choose a lower dose level as the RP2D, depending on toxicity considerations, dose reduction on subsequent cycles, and other considerations.
Time Frame: From initial study treatment to two cycles of study treatment
Measure: Number; unit: mg
Groups:
- Treatment (Vorinostat, Pembrolizumab): Patients receive vorinostat PO BID on days 1-5 and 8-12 and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Vorinostat, Pembrolizumab)
Number analyzed (Participants) | 52
mg | 200

3. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: The dose-limiting toxicity (DLT) observation period was 42 days (2 cycles). DLT assessment occurred on cycle 3, day 1 prior to receipt of cycle 3, day 1 of study therapy. Toxicities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03).
Time Frame: From initial study treatment to two cycles of study treatment, up to 42 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat 100mg + Pembrolizumab 200mg | Vorinostat 200mg + Pembrolizumab 200mg
Number analyzed (Participants) | 6 | 46
Participants | 1 | 1

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was calculated as the proportion of evaluable patients that had confirmed complete response (CR) or partial response (PR), as defined according to the 2014 Lugano Classification, exact 95% confidence intervals were calculated for these estimates.
Time Frame: From initial study treatment up to 36 21-day cycles
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vorinostat 100mg + Pembrolizumab 200mg | Vorinostat 200mg + Pembrolizumab 200mg
Number analyzed (Participants) | 6 | 46
percentage of participants | 50 [12 to 88] | 61 [45 to 75]

5. Secondary Outcome: Complete Response Rate (CR)
Description: CR was calculated as the proportion of evaluable patients that had confirmed complete response, as defined according to the 2014 Lugano Classification, exact 95% confidence intervals were calculated for these estimates.
Time Frame: From the initial treatment to 36 21-day cycles.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vorinostat 100mg + Pembrolizumab 200mg | Vorinostat 200mg + Pembrolizumab 200mg
Number analyzed (Participants) | 6 | 46
percentage of participants | 17 [0.4 to 64] | 35 [21 to 50]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored/assessed at each 21-day cycle treatment and up to 30 days post-last dose (up to 25 months) for AE or 90 days post-last dose (up to 27 months) for SAE. All-Cause Mortality was monitored/assessed up to 57 months post-treatment.
Arm/Group | Vorinostat 100mg + Pembrolizumab 200mg | Vorinostat 200mg + Pembrolizumab 200mg
All-Cause Mortality (participants affected / at risk) | 1/6 | 16/46
Serious Adverse Events (participants affected / at risk) | 1/6 | 8/46
Other Adverse Events (participants affected / at risk) | 6/6 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 100mg + Pembrolizumab 200mg (N=6) | Vorinostat 200mg + Pembrolizumab 200mg (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 100mg + Pembrolizumab 200mg (N=6) | Vorinostat 200mg + Pembrolizumab 200mg (N=46)
ANEMIA (Blood and lymphatic system disorders) | 2 (5) | 24 (66)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1) | 6 (10)
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 3 (4) | 16 (37)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (3) | 19 (39)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1)
MIDDLE EAR INFLAMMATION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 2 (2)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 6 (7)
BLEPHARITIS (Eye disorders) | 0 (0) | 1 (1)
BLURRED VISION (Eye disorders) | 0 (0) | 2 (3)
DRY EYE (Eye disorders) | 1 (1) | 3 (5)
EYE PAIN (Eye disorders) | 0 (0) | 2 (2)
FLASHING LIGHTS (Eye disorders) | 0 (0) | 1 (1)
WATERING EYES (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (3) | 24 (93)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOATING (Gastrointestinal disorders) | 0 (0) | 4 (4)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 14 (22)
DIARRHEA (Gastrointestinal disorders) | 2 (3) | 27 (126)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 6 (8)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 9 (10)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (8)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (3) | 4 (4)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (2) | 0 (0)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (2) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 34 (114)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 5 (7)
SALIVARY DUCT INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 20 (35)
CHILLS (General disorders) | 1 (1) | 7 (10)
EDEMA LIMBS (General disorders) | 1 (1) | 2 (2)
FATIGUE (General disorders) | 3 (4) | 31 (115)
FEVER (General disorders) | 0 (0) | 9 (20)
FINGER TIP PAIN (General disorders) | 0 (0) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 2 (2)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1)
HANDS SWOLLEN (General disorders) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 0 (0) | 2 (2)
INJECTION SITE REACTION (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 6 (10)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 7 (16)
PAIN (General disorders) | 0 (0) | 11 (11)
SWOLLEN HANDS (General disorders) | 0 (0) | 1 (3)
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
COMMON COLD (Infections and infestations) | 0 (0) | 1 (1)
CORONAVIRUS: HKU1 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4)
LUNG INFECTION (Infections and infestations) | 0 (0) | 3 (3)
PAPULOPUSTULAR RASH (Infections and infestations) | 0 (0) | 4 (7)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 7 (8)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 8 (12)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 10 (13)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 4 (9)
CARDIAC TROPONIN I INCREASED (Investigations) | 0 (0) | 2 (2)
CHOLESTEROL HIGH (Investigations) | 0 (0) | 1 (1)
CREATININE INCREASED (Investigations) | 1 (1) | 12 (23)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 0 (0) | 5 (7)
LYMPHOCYTE COUNT DECREASED (Investigations) | 6 (8) | 9 (29)
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (4) | 19 (69)
PLATELET COUNT DECREASED (Investigations) | 1 (3) | 20 (62)
WEIGHT GAIN (Investigations) | 1 (2) | 18 (41)
WEIGHT LOSS (Investigations) | 1 (1) | 18 (39)
WHITE BLOOD CELL DECREASED (Investigations) | 5 (7) | 20 (75)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 16 (26)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 4 (6)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 5 (9)
HYPERKALEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (6)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 8 (12)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 (2) | 9 (18)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (2) | 15 (23)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 14 (21)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2) | 25 (66)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1) | 17 (49)
OBESITY (Metabolism and nutrition disorders) | 1 (5) | 10 (22)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (15)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (9)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 13 (45)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (15)
DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
POLYPS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 11 (46)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 5 (11)
HEADACHE (Nervous system disorders) | 0 (0) | 13 (47)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
PARESTHESIA (Nervous system disorders) | 0 (0) | 4 (6)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 13 (28)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 4 (4)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 10 (15)
CONFUSION (Psychiatric disorders) | 0 (0) | 2 (2)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
HALLUCINATIONS (Psychiatric disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 12 (12)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 1 (11)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 3 (4)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 3 (3)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 5 (5)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
URINE DISCOLORATION (Renal and urinary disorders) | 0 (0) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
IRREGULAR MENSTRUATION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ALLERGIES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 20 (28)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (15)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (9)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (13)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (14)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (2) | 13 (23)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
WART (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 0 (0) | 2 (2)
HOT FLASHES (Vascular disorders) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 5 (10) | 41 (199)
HYPOTENSION (Vascular disorders) | 1 (1) | 15 (25)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT03150329/Prot_SAP_000.pdf